CLINICAL TRIAL: NCT04294901
Title: Engaging Patients to Promote Deprescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 18-228
Record Dates: First submitted 2020-02-24; First posted 2020-03-04 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Medical Overuse; Inappropriate Prescribing; Deprescriptions
Keywords: Physician-Patient Relations; Implementation Science; Decision Making, Shared

STUDY DESIGN:
Intervention Model Description: The investigators will target Veterans at three primary care sites who meet eligibility criteria for one of the PIM cohorts and are prescribed the target medication at the time of their scheduled primary care visit. Each PCP was assigned to receive three medication groups (i.e., PPIs, diabetes medications, and gabapentin) in a randomized order, and during each period of time for each medication/medication group assignment, prescriptions for that specific medication/medication group were assessed. Patients that received the specific medication or medication group from the PCP during the time of assignment were enrolled in the study. The study will begin with a 13-month retrospective baseline period, with one month for baseline subject identification and 12 months for observation of baseline subjects' deprescribing outcomes. The primary comparisons are between "brochure-intervention" patients and "baseline" patients (matched in terms of eligibility) from the same provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Patients prescribed gabapentin with a total daily dose >1800mg meeting inclusion/exclusion criteria who have a primary care appointment with a provider in the Gaba cohort; Patients prescribed either insulin or a sulfonylurea meeting inclusion/exclusion criteria who have a primary care appointment with a provider in the DM cohort; Patients prescribed a PPI meeting inclusion/exclusion criteria who have a primary care appointment with a provider in the PPI cohort
  Interventions: Behavioral: Direct to patient medication brochure
- Control (No Intervention): Historical control patients seen by intervention PCPs in the 18-12 months prior to the intervention window.

INTERVENTIONS:
Behavioral: Direct to patient medication brochure — An EMPOWER medication brochure, adapted to the VA, designed to educate and activate patients. These brochures provide detailed medication information, allow self-testing of indications for use, prompt reflection of experiences with potential side effects, discuss alternative therapies (medication and non-pharmacologic options), and provide a vignette of a patient who successfully stopped the medicine. They were designed for a 6th grade reading level and were based upon theories of patient activation, adult learning, and cognitive dissonance. The visually appealing brochure repeatedly emphasizes that patients should not make any medication changes without first consulting their health care providers.
  Arms: Intervention

SUMMARY:
One mechanism to reduce potentially inappropriate medications is through deprescribing, a deimplementation-based approach to thoughtfully discontinue a medication a patient is currently prescribed. Many interventions to overcome deprescribing barriers target the provider, who is already overburdened. Although some believe providers have primary responsibility for deprescribing, patient-initiated discontinuation discussions can effectively facilitate deprescribing. In a single-site pilot study, the investigators successfully engaged VA Primary Care patients to facilitate deprescribing of select potentially inappropriate medications. The investigators now propose a multisite randomized controlled trial of engaging Veterans who may be deprescribing candidates. By study end, the investigators will have established the effectiveness of an innovative, low-tech, patient-focused intervention to promote deprescribing, thereby directly improving quality, safety, and value of VA care while also setting the stage for generalization of this approach to other potentially inappropriate medications.

DETAILED DESCRIPTION:
Background - Despite multiple provider- and system-level interventions to reduce potentially inappropriate medications (PIMs), many Veterans are still prescribed drugs that provide little benefit, placing them at unnecessary risk of adverse drug events (ADEs). One mechanism to reduce PIMs is through deprescribing, a de-implementation-based approach to thoughtfully discontinue a medication a patient is currently prescribed.

Many Choosing Wisely recommendations address PIMs. Specifically, proton pump inhibitors (PPIs), a medicine used to reduce gastric acid, should be de-escalated to the lowest dose necessary to provide relief. Many older patients with diabetes are over-controlled, with blood sugar levels lower than recommended, yet remain on multiple diabetes medicines and may be able to use fewer medicines. These patients are also at higher risk of low blood sugar from insulin and sulfonylureas, and should have limited use of these agents.

Finally, gabapentin is often used off-label to treat pain, with greatly increased use over the past several years. There are many barriers to deprescribing PIMs. Many interventions solely target the prescribing provider. Although some believe providers have primary responsibility for deprescribing, patient initiation of discontinuation conversations can effectively facilitate deprescribing. In a single-site pilot study, the investigators successfully reduced PIMs by engaging VA Primary Care patients by providing them with Veteran-centric EMPOWER ("Eliminating Medications through Patient Ownership of End Results") brochures. However, it is not known if this approach will be as successful for Veterans with other chronic conditions or at non-pilot sites.

Aims - The investigators propose three aims. 1) Examine the impact of a patient-centered intervention to change provider prescribing (the primary outcome), as determined by the frequency with which medications are either deprescribed or de-escalated. 2) Examine the effect of a patient-centered intervention on engaging patients, via post-visit surveys of Veterans' interaction with the brochures and their influence on deprescribing discussions and deprescribing. 3) Using qualitative methods, identify key organizational contextual factors related to intervention fidelity, feasibility, acceptability, and appropriateness to support future implementation.

Methods and Innovation - The investigators propose a multisite quasi-experimental trial using a Hybrid Type I Effectiveness-Implementation design of providing EMPOWER brochures directly to Veterans who may be deprescribing candidates for three cohorts of PIMs (PPIs, diabetes medications, and gabapentin). The investigators will mail brochures in advance of scheduled primary care visits, unlike distribution methods used in other studies. The primary outcome will be the composite of deprescribing and de-escalation of target medications, identified in pharmacy dispensing records of the Corporate Data Warehouse (Aim 1). Mail-based surveys sent after the scheduled primary care visit will assess patient engagement with the brochure and its impact on patient-provider communication (Aim 2). Finally, qualitative data from clinicians and staff addressing Proctor's Implementation Outcomes will provide the foundation for future implementation strategies (Aim 3).

Significance and Next Steps - The study directly addresses multiple Veteran Care Priorities, including health care value, primary care practice, quality/safety, and Whole Health, and is aligned with current VA initiatives to prioritize patient preferences via individually-tailored, proactive care plans. The proposed work is strongly supported by Pharmacy Benefits Management and Office of Patient Centered Care and Cultural Transformation, which will facilitate the dissemination of findings to improve the quality and safety of medication use within VA. By study end, the investigators will have established the effectiveness of an innovative, low-tech, patient-focused intervention to promote deprescribing of commonly used medications for three populations, thereby directly improving quality, safety, and value of VA care while also setting the stage for wider implementation and generalization of this approach to other potentially inappropriate medications.

ELIGIBILITY:
Inclusion Criteria:

* Veteran with a Primary Care appointment at one of three Veteran Affairs Medical Centers (including Community Based Outpatient Clinics)

  * PPI Cohort:

    * >90 consecutive days of PPI at any dose
  * Diabetes Cohorts:

    * HbA1c <7%
    * At least one of Age >65 years
    * Renal impairment
    * Cognitive impairment
    * either >90 consecutive days insulin or sulfonylurea or >90 consecutive days of >2 DM medications (neither of which is insulin or sulfonylurea)
  * Gaba Cohort:

    * >90 consecutive days with total daily dose >1800mg

Exclusion Criteria:

* PPI Cohort Exclusions:

  * Diagnosis warranting PPI treatment
  * Medication warranting PPI treatment
* Gaba Cohort Exclusions:

  * Neuropathic pain
  * Seizure disorder
  * and/or Cancer-related pain

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5946 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-10-07 (Actual); Study Completion 2023-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Linsky, MD MSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (4):
- United States (4):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Central Western Massachusetts Healthcare System, Leeds, MA, Leeds, Massachusetts
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
Datasets meeting VA standards for disclosure to the public will be made available within 1 year of publication. Prior to distribution, a local privacy officer will certify that all datasets contains no PHI. Final data sets will be maintained locally until enterprise-level resources become available for long-term storage and access. Guidance on request and distribution processes will be provided by ORD. Those requesting data will be asked to sign a Letter of Agreement.
Time Frame: Within 1 year of publication
Access Criteria: Those requesting data will be asked to sign a Letter of Agreement.

REFERENCES:
- [Background] Zimmerman KM, Linsky AM. A narrative review of updates in deprescribing research. J Am Geriatr Soc. 2021 Sep;69(9):2619-2624. doi: 10.1111/jgs.17273. Epub 2021 May 15. PMID 33991423
- [Background] Niznik JD, Zhao X, Slieanu F, Mor MK, Aspinall SL, Gellad WF, Ersek M, Hickson RP, Springer SP, Schleiden LJ, Hanlon JT, Thorpe JM, Thorpe CT. Effect of Deintensifying Diabetes Medications on Negative Events in Older Veteran Nursing Home Residents. Diabetes Care. 2022 Jul 7;45(7):1558-1567. doi: 10.2337/dc21-2116. PMID 35621712
- [Derived] Jones KF, Stolzmann K, Wormwood J, Pendergast J, Miller CJ, Still M, Bokhour BG, Hanlon J, Simon SR, Rosen AK, Linsky AM. Effectiveness of Patient-Directed Education to Sustain Deprescribing: A Pragmatic Trial. Drugs Aging. 2025 Nov;42(11):1073-1083. doi: 10.1007/s40266-025-01251-z. Epub 2025 Oct 18. PMID 41108442

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Patients who received an EMPOWER brochure two weeks before their primary care appointment.
  Direct to patient medication brochure: An EMPOWER medication brochure, adapted to the VA, designed to educate and activate patients. These brochures provide detailed medication information, allow self-testing of indications for use, prompt reflection of experiences with potential side effects, discuss alternative therapies (medication and non-pharmacologic options), and provide a vignette of a patient who successfully stopped the medicine. They were designed for a 6th grade reading level and were based upon theories of patient activation, adult learning, and cognitive dissonance. The visually appealing brochure repeatedly emphasizes that patients should not make any medication changes without first consulting their health care providers.
- Historical Control Group: The historical control cohort were seen by the same PCPs at the same sites as our intervention cohort from October 2019 to April 2020 (eighteen months to one year before the intervention timeframe).
  The PPI group included adult patients of any age with an active prescription for any PPI with at least 90 consecutive days on the medication in the prior year, excluding diagnoses for which PPI continuation would be appropriate (e.g., Barrett's esophagus, or those prescribed chronic anti-inflammatory drugs associated with peptic ulcers).
  The Gabapentin group included adult patients of any age with an active prescription of gabapentin >1800mg/day with at least 90 consecutive days on the medication in the prior year, excluding patients with potential indications for use, including neuropathic pain, seizure disorders, and cancer-related pain.
  The hypoglycemia-risk group included patients with diabetes based upon ICD-10-CM diagnosis codes, most recent HbA1c <7%, as well as one or more of the following criteria: 1) age 65 years or older, 2) renal insufficiency defined as creatinine >2 mg/dL, and/or 3) a diagnosis of cognitive impairment or prescription for an acetylcholinesterase inhibitor (e.g., donepezil). Patients in the hypoglycemia-risk group had an active prescription for insulin or sulfonylurea with at least 90 consecutive days on the medication in the prior year.
Period: Overall Study
Arm/Group | Intervention Group | Historical Control Group
Started | 3206 | 2740
PPI (These are the subjects in the PPI medication group who completed the study.) | 2064 | 2000
DM-Hypoglycemia Risk (These are the subjects in the DM-Hypoglycemia medication group who completed the study.) | 378 | 427
Gabapentin (These are the subjects in the Gabapentin medication group who completed the study.) | 97 | 105
Completed | 2539 | 2532
Not Completed | 667 | 208
Not completed — Death | 86 | 110
Not completed — Provider did not have historical control patients | 581 | 0
Not completed — Provider did not have intervention patients | 0 | 98

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Historical Control Group | Total
Number analyzed (Participants) | 3206 | 2740 | 5946
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.15 (12.03) | 70.61 (12.59) | 70.68 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 141 | 336
  Male | 3011 | 2599 | 5610
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2287 | 2029 | 4316
  Black | 459 | 297 | 756
  American Indian or Alaskan Native | 42 | 36 | 78
  Asian | 36 | 53 | 89
  Native Hawaiian or Pacific Islander | 27 | 33 | 60
  Missing | 355 | 292 | 647
Medication Group [Count of Participants; unit: Participants]
  Proton Pump Inhibitor | 2624 | 2157 | 4781
  Gabapentin | 121 | 112 | 233
  Hypoglycemic | 461 | 471 | 932

OUTCOME MEASURES:

1. Primary Outcome: Deprescribing
Description: Non-refill of the medication in the 6 months following the primary care appointment (i.e., cessation) or any reduction in the total daily dose (i.e., de-escalation). There is an exception to the de-escalation rule for insulin, where only complete cessation will qualify since dose changes are less likely to be reflected in the order compared to oral medications.
Time Frame: 6 months post-index date
Population: It is pre-specified in the Study Protocol and Statistical Analysis Plan to assess all medication groups combined within the Intervention and Control Arms/Groups
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Group: Patients who received an EMPOWER brochure two weeks before scheduled primary care appointments.
  Direct to patient medication brochure: An EMPOWER medication brochure, adapted to the VA, designed to educate and activate patients. These brochures provide detailed medication information, allow self-testing of indications for use, prompt reflection of experiences with potential side effects, discuss alternative therapies (medication and non-pharmacologic options), and provide a vignette of a patient who successfully stopped the medicine. They were designed for a 6th grade reading level and were based upon theories of patient activation, adult learning, and cognitive dissonance. The visually appealing brochure repeatedly emphasizes that patients should not make any medication changes without first consulting their health care providers.
Arm/Group | Intervention Group | Historical Control Group
Number analyzed (Participants) | 2539 | 2532
Participants | 748 | 653
Statistical Analysis 1: Comparison: Intervention Group vs Historical Control Group; It is pre-specified in the Study Protocol and Statistical Analysis Plan to assess all medication groups combined within the Intervention and Control Arms/Groups; Test type: Superiority; p = 0.008, Mixed Models Analysis; Binary mixed effect model with patients nested in providers nested in facilities; Odds Ratio (OR) = 1.21, 95% CI 2-sided [1.05 to 1.38]

2. Secondary Outcome: Deprescribing Conversations
Description: Patient report of a conversation about deprescribing during the index primary care visit. Note that this Outcome Measure was only assessed in a subsample of the "Intervention Group" Arm/Group participants and not at all in the "Historical Control Group" Arm/Group subjects.
Time Frame: Index visit until survey completion (up to 8 weeks post-index visit)
Population: Note that this Outcome Measure was only assessed in a subsample of the "Intervention Group" Arm/Group participants who responded to the survey. It was not assessed at all in the "Historical Control Group" Arm/Group subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Gabapentin (Gaba): Patients prescribed gabapentin with a total daily dose >1800mg without exclusion criteria who have a primary care appointment with a provider in the Gaba cohort
  Direct to patient medication brochure: An EMPOWER medication brochure, adapted to the VA, designed to educate and activate patients. These brochures provide detailed medication information, allow self-testing of indications for use, prompt reflection of experiences with potential side effects, discuss alternative therapies (medication and non-pharmacologic options), and provide a vignette of a patient who successfully stopped the medicine. They were designed for a 6th grade reading level and were based upon theories of patient activation, adult learning, and cognitive dissonance. The visually appealing brochure repeatedly emphasizes that patients should not make any medication changes without first consulting their health care providers.
- Diabetes (DM): Patients prescribed either insulin or a sulfonylurea meeting inclusion/exclusion criteria who have a primary care appointment with a provider in the DM cohort
  Direct to patient medication brochure: An EMPOWER medication brochure, adapted to the VA, designed to educate and activate patients. These brochures provide detailed medication information, allow self-testing of indications for use, prompt reflection of experiences with potential side effects, discuss alternative therapies (medication and non-pharmacologic options), and provide a vignette of a patient who successfully stopped the medicine. They were designed for a 6th grade reading level and were based upon theories of patient activation, adult learning, and cognitive dissonance. The visually appealing brochure repeatedly emphasizes that patients should not make any medication changes without first consulting their health care providers.
- Proton Pump Inhibitor (PPI): Patients prescribed a PPI meeting inclusion/exclusion criteria who have a primary care appointment with a provider in the PPI cohort
  Direct to patient medication brochure: An EMPOWER medication brochure, adapted to the VA, designed to educate and activate patients. These brochures provide detailed medication information, allow self-testing of indications for use, prompt reflection of experiences with potential side effects, discuss alternative therapies (medication and non-pharmacologic options), and provide a vignette of a patient who successfully stopped the medicine. They were designed for a 6th grade reading level and were based upon theories of patient activation, adult learning, and cognitive dissonance. The visually appealing brochure repeatedly emphasizes that patients should not make any medication changes without first consulting their health care providers.
Arm/Group | Gabapentin (Gaba) | Diabetes (DM) | Proton Pump Inhibitor (PPI)
Number analyzed (Participants) | 40 | 226 | 1116
Participants | 12 | 37 | 353

ADVERSE EVENTS:
Time Frame: Potential medication-specific adverse drug withdrawal events (ADWEs) within 12 months after index date.
Description: All participants that started the study were assessed for All-Cause Mortality. Only the Safety Analysis Population was assessed for Serious and Other Adverse Events ADWEs - a priori specified serious adverse drug withdrawal events: upper gastrointestinal bleed for PPIs, diabetic ketoacidosis or hyperosmolar hyperglycemic state for insulin and sulfonylureas, and seizure for gabapentin. It was pre-specified to combine all medication groups within the Intervention and Control Arms/Groups.
Arm/Group | Intervention Group | Historical Control Group
All-Cause Mortality (participants affected / at risk) | 86/3206 | 110/2740
Serious Adverse Events (participants affected / at risk) | 25/2539 | 26/2532
Other Adverse Events (participants affected / at risk) | 0/2539 | 0/2532
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=2539) | Historical Control Group (N=2532)
Potential adverse drug withdrawal event (General disorders) | 25 (25) | 26 (26) — upper gastrointestinal bleed for proton pump inhibitors (PPIs), diabetic ketoacidosis or hyperosmolar hyperglycemic state for insulin and sulfonylureas, and seizure for gabapentin.

LIMITATIONS AND CAVEATS:
Total numbers for Baseline Characteristics are less than the number of subjects due to missing data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT04294901/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT04294901/SAP_001.pdf